CLINICAL TRIAL: NCT06149897
Title: Feasibility and Effectiveness of Tdcs in a Multimodal Treatment With Health Education and Aerobic Exercise in the Treatment of Post-stroke Fatigue.
Brief Title: Feasibility and Effectiveness of tDCS in the Treatment of Post-stroke Fatigue (EFECTS).
Acronym: EFECTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Inés García Bouyssou, Physical therapist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCB/2022/1193
Record Dates: First submitted 2023-11-14; First posted 2023-11-29 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: tdcs; post stroke fatigue
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): * Therapeutic education about post-stroke fatigue
  * Sham stimulation with tDCS: Anode placed in F3 and cathode in O2, 20 minutes.
  * Aerobic exercise measured with Borg scale (moderate intensity)
  Interventions: Device: tDCS
- Experimental group (Active Comparator): * Therapeutic education about post-stroke fatigue
  * Stimulation with tDCS: Anode placed in F3 and cathode in O2, intensity 2mA during 20 minutes.
  * Aerobic exercise measured with Borg scale (moderate intensity)
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Non invasive brain stimulation with sham and active comparators
  Other Names: physical exercise; therapeutic education

SUMMARY:
This study aims to analyze the use of non-invasive brain stimulation (tDCS) is beneficial for the treatment of post-stroke fatigue.

DETAILED DESCRIPTION:
A single-blind randomized clinical trial will be conducted. The intervention will consist of 8 20-minute tDCS sessions conducted over four weeks. The stimulation will be performed by applying the stimulation to the dorsolateral prefrontal cortex on the left side (F3) and the cathode will be at point O2 of the right hemisphere. The study will consist of two groups: the control group in which sham stimulation will be applied and therapeutic education and aerobic exercise; the intervention group in which stimulation, therapeutic education and therapeutic exercise will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* First stroke within 45 (+-7) days of the ischemic or hemorrhagic episode.
* Ability to understand and execute simple instructions
* Over 18 years.
* Fatigue Scale of fatigue severity with a score greater than or equal to 24

Exclusion Criteria:

* A score > 2 on the modified Rankin Scale (mRS) before the stroke.
* Patients with decompensated cardiorespiratory and/or psychiatric pathology.
* Comorbidity causing disproportionate fatigue, such as long-term COVID.
* Patients who are cancer survivors or who are undergoing cancer treatment.
* Patients with a history of epilepsy or who are taking antiepileptic medication.
* Patents with major depression.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Fatigue Assessment Scale | Baseline, 1 month post intervention and 3 months post intervention. Reported through study completion, an average of 1 year.
  The scale consists of 10 questions about the characteristics of fatigue in the current daily routine, which are rated on a five-point range from 1, "never," to 5, "always." Higher scores indicate more fatigue, with a cut-off point of ≥24 defining the presence of fatigue.
HADS | Baseline, 1 month post intervention and 3 months post intervention. Reported through study completion, an average of 1 year.
  It is a scale that can be used both at the hospital and outpatient level. It consists of 14 questions: 7 questions related to depression and another 7 related to anxiety. An independent score on each scale of ≥ 8 will be suggestive of depression and/or anxiety.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale | Baseline. Reported through study completion, an average of 1 year.
  It is a scale with 15 items that is used to measure the severity of stroke. It includes different areas: level of consciousness, eye movements, integrity of visual fields, facial movements, muscle strength, sensitivity, coordination, language and negligence. Each item is scored on an ordinal scale from 0 to 2, 0 to 3 or 0 to 4. The total is added and a score is obtained that can range from 0 to 42, the higher the score, the greater the deficits.
Borg Modified Scale | During the sessions. Reported through study completion, an average of 1 year.
  The Borg scale is a tool that measures a person's perception of exertion, shortness of breath, and fatigue during physical exertion. It is a modified scale, it is an 11-point scale that ranges from 0=no fatigue to 10=very great effort.
PROMIS-Sleep | Baseline, 1 month post intervention and 3 months post intervention. Reported through study completion, an average of 1 year.
  This is a Likert-type scale that evaluates the quality of sleep during the last week. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Modified Rankin Scale | Baseline, 1 month post intervention and 6 months post intervention. Reported through study completion, an average of 1 year.
  It is the most commonly used functional measure in stroke research, particularly in studies evaluating the effectiveness of treatments. The scale is numerical and ranges from 0 to 6. 0: no symptoms; 1: without significant disability (the patient is able to carry out his/her usual activities and obligations); 2: mild disability; 3: moderate disability; 4: moderately severe disability; 5: severe disability (totally dependent patient); 6: death.
International Physical Activity Questionnaire (IPAQ) | Baseline, 1 month post intervention and 3 months post intervention. Reported through study completion, an average of 1 year.
  To measure the level of physical activity during the last week. There are two forms of output from scoring the IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity. A MET is a multiple of your estimated resting energy expenditure. One MET is what you expend when you are at rest. Therefore 2 METS is twice what you expend at rest. To get a continuous variable score from the IPAQ (MET minutes a week) we will consider walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS.
Eq-5D | Baseline, 1 month post intervention and 3 months post intervention. Reported through study completion, an average of 1 year.
  Assess the quality of life perceived by the patients. The scale ranges from 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state' or 'the worst health you can imagine'). This is used to obtain a respondent's stated preference values, not to record their own health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain, Spain